CLINICAL TRIAL: NCT07383402
Title: The Efficacy of Intra-sinus Povidone-iodine/Budesonide Gel Forming Suspension Following Endoscopic Sinus Surgery for Chronic Rhinosinusitis: a Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Intra-Sinus Povidone-Iodine and Budesonide After Endoscopic Sinus Surgery for Chronic Rhinosinusitis
Acronym: PVP-I
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amin Javer (Other)
Responsible Party: Sponsor-Investigator, Amin Javer, MD, St. Paul's Hospital, Canada
Organization: St. Paul's Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H24-02473
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Rhinosinusitis (CRS)
Keywords: Povidone Iodine; Budesonide
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone-Iodine and Budesonide Gel-Forming Suspension (Active Comparator): Participants randomized to this arm will receive an intra-sinus gel-forming suspension containing povidone-iodine and budesonide administered at the completion of endoscopic sinus surgery.
  Interventions: Drug: Povidone-Iodine and Budesonide Gel-Forming Suspension
- Placebo Gel-Forming Suspension (Placebo Comparator): Participants randomized to this arm will receive an intra-sinus placebo gel-forming suspension without active drug administered at the completion of endoscopic sinus surgery.
  Interventions: Drug: Placebo Gel-Forming Suspension

INTERVENTIONS:
Drug: Povidone-Iodine and Budesonide Gel-Forming Suspension — A gel-forming suspension containing povidone-iodine and budesonide administered intra-sinus at the completion of endoscopic sinus surgery, intended to reduce postoperative inflammation and improve sinus cavity healing.
  Arms: Povidone-Iodine and Budesonide Gel-Forming Suspension
Drug: Placebo Gel-Forming Suspension — A gel-forming suspension without povidone-iodine or budesonide administered intra-sinus at the completion of endoscopic sinus surgery.
  Arms: Placebo Gel-Forming Suspension

SUMMARY:
Endoscopic sinus surgery (ESS) is commonly performed in patients with chronic rhinosinusitis (CRS) to improve sinus drainage and allow better delivery of topical therapies after surgery. Despite surgery, postoperative inflammation can persist and negatively affect healing and outcomes.

This randomized, double-blind, placebo-controlled clinical trial will evaluate whether intra-sinus administration of a gel-forming suspension containing povidone-iodine and budesonide improves postoperative endoscopic outcomes of the sinus cavities three months following ESS, compared with placebo.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a chronic inflammatory condition that can significantly impact quality of life. Endoscopic sinus surgery (ESS) is performed in patients with CRS who do not respond adequately to medical therapy, with the goals of improving sinus drainage, reducing disease burden, and facilitating postoperative topical treatment delivery. However, postoperative inflammation and impaired mucosal healing may persist despite surgery and standard postoperative care.

Povidone-iodine (PVP-I) has broad antimicrobial and anti-inflammatory properties, while budesonide is a corticosteroid commonly used intranasally to reduce sinonasal inflammation. Although both agents are individually used in sinonasal care, the efficacy and safety of their combined intra-sinus administration in a gel-forming suspension following ESS have not been well established.

This randomized, double-blind, placebo-controlled clinical trial will evaluate the efficacy and safety of an intra-sinus gel-forming suspension containing PVP-I and budesonide administered at the time of ESS in adult patients with CRS. Participants will be randomized to receive either the investigational gel-forming suspension or a placebo gel following completion of surgery.

Participants will be followed postoperatively according to standard clinical care. The primary outcome will assess endoscopic appearance of the sinus cavities three months following ESS using a validated endoscopic scoring system. Secondary outcomes will evaluate postoperative sinonasal symptoms, mucosal healing, and treatment-related adverse events.

The results of this study will help determine whether intra-sinus delivery of a combined PVP-I and budesonide gel-forming suspension improves postoperative endoscopic outcomes and supports its use as an adjunctive therapy following ESS in patients with CRS.

ELIGIBILITY:
Inclusion Criteria:

Age 19 years or older Scheduled for Endoscopic Sinus Surgery (ESS)

Exclusion Criteria:

Cystic fibrosis Systemic vasculitis Known or suspected hypersensitivity to povidone iodine Inhaled drug use (i.e., cocaine) in the preceding 6 months Nasal tumors Known or suspected immunodeficiencies Pregnant women Breast feeding women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Lund-Kennedy (MLK) Endoscopic Score | 12 weeks postoperatively
  Change in the Modified Lund-Kennedy (MLK) endoscopic score comparing baseline to 12 weeks following endoscopic sinus surgery. The MLK score is a validated endoscopic scoring system assessing sinonasal inflammation, including edema and polyps, with higher scores indicating worse disease severity.

SECONDARY OUTCOMES:
Scar Tissue Formation | Up to 24 weeks postoperatively
  Presence and severity of postoperative scar tissue formation assessed by nasal endoscopy.

IPD SHARING:
Plan to Share IPD: Undecided